CLINICAL TRIAL: NCT07370818
Title: An Open-label, Dose-finding and Randomized Active-controlled, Phase 2 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of JPI-547 With Bevacizumab Maintenance Therapy in Relapsed Ovarian Cancer Patients Previously Treated With PARP Inhibitor Maintenance Therapy and Responding to Last Platinum Chemotherapy
Brief Title: To Evaluate the Efficacy and Safety of JPI-547 in Combination With Bevacizumab as Maintenance Therapy in Relapsed Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPI-547-202
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JPI-547+Bevacizumab (Experimental)
  Interventions: Drug: JPI-547; Drug: Bevacizumab
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: JPI-547 — taking JPI-547
  Arms: JPI-547+Bevacizumab
Drug: Bevacizumab — administration Bevacizumab

SUMMARY:
This study aims to to evaluate the efficacy, safety, and pharmacokinetics of JPI- 547 with bevacizumab maintenance therapy in relapsed ovarian cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent ovarian cancer, fallopian tube cancer, or primary peritoneal cancer [High-grade serous carcinoma (HGSC), Grade 2/3 endometrioid carcinoma]
* Patients whose BRCA 1/2 gene mutation status and/or Homologous Recombination Deficiency (HRD) status.
* Patients who received platinum-based chemotherapy followed by PARP inhibitor maintenance therapy,
* Patients who had received chemotherapy before participating in the clinical trial and responded to platinum-based chemotherapy.
* Those with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Individuals with confirmed adequate hematological, renal, and hepatic function (laboratory tests may be repeated once during the screening period)

Exclusion Criteria:

* Patients with a history of severe drug hypersensitivity or hypersensitivity to the investigational drug, its components, or drugs within the same class.
* Individuals with dysphagia
* Patients with a confirmed specific medical history or a past surgical history.
* Patients with specific comorbidities or medical abnormalities.
* Pregnant women, lactating women, or women of childbearing potential who do not agree to use appropriate contraception during the clinical trial period and for 24 weeks after administration of the investigational medicinal product.
* Those who have administered other investigational products or have received investigational medical device procedures within 4 weeks of the baseline
* Other patients who are inappropriate or unable to participate in this clinical study at the discretion of the investigator.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum tolerated dose (MTD) and recommended dose (RD)(RP2D) | The dose-limiting toxicity evaluation window is 21 days
Part B: Progression free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 74 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes